CLINICAL TRIAL: NCT02729376
Title: An Open-Label, Single-Dose Study to Assess the Absorption, Metabolism, Excretion, and Mass Balance of Radiolabeled Galeterone in Healthy Male Subjects After Oral Administration
Brief Title: Single-Dose Study to Assess the Absorption, Metabolism, Excretion, and Mass Balance of Radiolabeled Galeterone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LTN PHARMACEUTICALS, INC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TOK-200-18
Record Dates: First submitted 2016-02-26; First posted 2016-04-06 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — 3-hydroxy-17-(1H-benzimidazole-1-yl)androsta-5,16-diene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single dose of [14C]-galeterone (Experimental): [14C]-galeterone will be supplied as 325 mg capsules (powder in capsule [PIC]). The treatment to be administered will be 2600 mg (~500 µCi) (8 x 325 mg capsules).
  Interventions: Drug: galeterone

INTERVENTIONS:
Drug: galeterone

SUMMARY:
This is an open label, single dose, 1 period study of [14C] galeterone.

DETAILED DESCRIPTION:
This is an open label, 1 period study under fed conditions. Six (6), healthy, adult, non tobacco using, male subjects will be enrolled. Screening of subjects will occur within 28 days prior to dosing. On Day 1, a single dose of radio-labeled galeterone will be administered orally. Blood, urine, and fecal samples will be collected until release criteria are met to measure total radioactivity, for analysis of galeterone concentrations, and for potential metabolic profiling.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male, 19 to 55 years of age, inclusive, at screening.
2. Continuous non smoker who has not used nicotine containing products for at least 3 months prior to dosing.
3. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

1. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI.
2. History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the subject by their participation in the study.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Radioactivity concentration equivalents in plasma | 168 hours
Single dose galeterone concentrations in plasma | 168 hours
Route(s) of elimination of a single [14C]galeterone dose | 8 days
Mass balance of a single [14C]galeterone dose | 8 days
Ratio of whole blood to plasma 14C radioactivity | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Karen J Ferrante, MD, Study Chair — Tokai Pharmaceuticals, Inc.
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No